CLINICAL TRIAL: NCT07159308
Title: Enhancing Motivation to Complete Daily Living Skills Among Transition-aged Autistic Youth
Brief Title: Motivation for Daily Living Skills
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-023525
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder (ASD); Motivation
Keywords: Interventions; Motivation; Autism Spectrum Disorder; Daily Living Skills; Transition to Adulthood; behavior therapy; motivational interviewing
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intrinsic Motivation Treatment (Experimental): Individuals assigned to this group will participate in the Intrinsic Motivation Treatment, which focuses on exploring a person's reasons for improving their completion of the daily living skill, such as reaching their goal of independence.
  Interventions: Behavioral: Intrinsic Motivation Treatment
- Extrinsic Motivation Treatment (Active Comparator): Individuals assigned to this group will participate in the Extrinsic Motivation Treatment. This treatment explores a person finding outside sources of motivation, such as treating themselves to something like or want.
  Interventions: Behavioral: Extrinsic Motivation Treatment
- Combined Intrinsic and Extrinsic Motivation Treatment (Experimental): Individuals assigned to this group will participate in the Combined Intrinsic and Extrinsic Motivation Treatment. This treatment combines methods from the Intrinsic Motivation Treatment and the Extrinsic Motivation Treatment. For example, exploring both a person's reasons behind wanting to improve upon their completion of a daily living skill as well as what outside sources will help increase their motivation to improve upon that skill.
  Interventions: Behavioral: Combined Intrinsic and Extrinsic Motivation Treatment

INTERVENTIONS:
Behavioral: Intrinsic Motivation Treatment — The Intrinsic Motivation treatment utilizes principles of Motivational Interviewing to help autistic young adults increase their desire and completion of daily living skills. This is a five-session intervention. Each clinical session is 60 minutes long. The goals of the treatment are to enhance motivation and behavior change.
  Arms: Intrinsic Motivation Treatment
Behavioral: Extrinsic Motivation Treatment — The Extrinsic Motivation treatment utilizes behavioral principles to help autistic adolescents and young adults create reward schedules and behavioral tracking sheets to enhance desire and completion of daily living skills. This is a five-session intervention. Each clinical session is 60 minutes long. The goals of the treatment are to enhance motivation and behavior change.
  Arms: Extrinsic Motivation Treatment
Behavioral: Combined Intrinsic and Extrinsic Motivation Treatment — The Combined Intrinsic and Extrinsic Motivation treatment combines elements of both intrinsic and extrinsic motivation treatments to enhance desire and completion of daily living skills. This is a five-session intervention. Each clinical session is 60-90 minutes long. The goals of the treatment are to enhance motivation and behavior change.
  Arms: Combined Intrinsic and Extrinsic Motivation Treatment

SUMMARY:
The goal of this clinical trial is to enhance motivation to complete daily living skills among 16 to 25-year-old autistic teens and young adults. Here are the main questions the trial aims to answer:

Can this trial improve motivation to complete daily living skills for skills that people know how to do but struggle to do them consistently?

Can this trial improve completion of the daily living skill that the participant identifies they want to do more often?

Do people report feeling more empowered to complete the daily living skill they want to do more often?

Are there any characteristics of a person that make them more or less likely to benefit from the treatment?

Researchers will compare treatments that target different types of motivation:

* One treatment focuses on internal motivation and explores what is important to someone and then connect that value back to their daily living skill goal.
* A second treatment focuses on external motivation and will explore a person finding outside sources of motivation, like rewards.
* A third treatment will use a combination of both methods.

Autistic teens and young adults enrolled in this study will also be asked to choose someone in their life to be involved in the study with them. This person is called an "Important Person" (IP) and can be anyone close to them, like a family member, friend, roommate, partner, etc. The IP will be expected to support the teen/young adult throughout this treatment.

Participants and their IPs will:

* Complete five 'talk' therapy sessions that will last 60 to 90 minutes. The IPs will join the last 15 minutes of each session)
* Be assigned to one of the three motivation treatments
* Fill out questionnaires before the first session, after sessions 2 through 5, and 2 weeks after therapy ends

DETAILED DESCRIPTION:
Many autistic teens and young adults often have a hard time doing the everyday skills they need to live on their own. These daily living skills (DLS) include things like taking care of themselves (like showering and getting dressed), doing chores at home (like cooking and cleaning), and handling things in the community (like saving money). Even if someone is able to do these skills, they might still struggle to do them. This shows that being able and knowing how to do these skills isn't the only important part-other things can make it hard to do daily tasks, like motivation.

Early research shows that some autistic young adults may not feel very motivated to do these daily tasks. There are different types of motivation. The researchers made three programs that focus on these different types.

One program focuses on intrinsic (internal) motivation and uses Motivational Interviewing strategies. Motivational Interviewing is a type of therapy that helps people find their personal reasons for making changes in their lives. This program will explore what is important to the participant and connect that value back to their daily living skill goal.

The researchers also made an extrinsic (external) motivation program. This program uses different behavioral strategies and will focus on a person finding outside sources of motivation. Some examples of these strategies are tracking how many times the participant completes their daily living skill in a week and giving themself a reward (like 'skin' in a video game or a t-shirt of their favorite band) if they reach their goal.

The third program is a combined program. This program includes activities from both the extrinsic motivation and intrinsic motivation programs explained above.

This study will compare these three programs in a preliminary efficacy trial. Preliminary efficacy means that this is the first trial where the researchers will look if there any benefits the participants may get from the treatments. The goal of this trial is to see which program helps autistic teens and young adults (ages 16-25) feel more motivated to do daily living skills. The results will help researchers plan a bigger study to find out whether intrinsic motivation, extrinsic motivation, or the combination of the two together work best.

The main questions the researchers of this trial want to answer are:

* Can the trial improve motivation to complete daily living skills for skills that people know how to do but struggle to do them consistently?
* Can the trial improve completion of the daily living skill that the participant identifies they want to do more often?
* Do people report feeling more empowered to complete the daily living skill they want to do more often?
* Are there any characteristics of a person that make them more or less likely to benefit from the treatment?

Another part of this treatment program is looking at social support. All teens/young adults enrolled in this study will be asked to choose someone in their life to be involved in the study with them. This person is called an 'Important Person' (IP) and can be anyone close to them, like a family member, friend, roommate, partner, etc. The IP will be expected to support the teen/young adult throughout this treatment.

All three programs have 5 therapy sessions and the follow-up session two weeks later. Sessions 1 through 5 includes answering some questionnaires and doing a 60-minute or 90-minute therapy session with a trained clinician. The IPs will join the last 15 minutes of each session and answer some questionnaires. These sessions will be in-person at the Children's Hospital of Philadelphia at their Philadelphia campus. The follow-up session includes both the teen/young adult participants and their IPs. This session can be done online and only involves answering some questionnaires. The goal of this session is to see if people stay motivated after the programs end.

Participation in this trial should not take more than 9 weeks and has three phases: a Screening and Consent Phase, Intervention Phase, and Follow-Up Phase.

In the Screening and Consent Phase, people who are interested will fill out a short form online to see if they are eligible to join this study. Then, they will have a follow-up call on Microsoft Teams with someone from the research team to confirm they are eligible and to collect their consent to join the study if they want to. After that, they get their study schedule and move into the Intervention Phase. The Intervention Phase includes the 5 therapy sessions that are part of the treatment programs and answering questionnaires. The trial ends with the Follow-Up phase where the participant and IP will receive a link to their final questionnaires two weeks after their last therapy session.

A possible benefit from participating in this study is that the treatments might help the teens/young adults feel more motivated to do daily living skills they want to do more often. They and their IP will also receive payment for completing the questionnaires.

ELIGIBILITY:
Inclusion Criteria for Autistic Teens and Young Adults:

* Age 16-25 years
* Participants reporting an autism diagnosis from a qualified provider (Psychiatrist, Psychologist, Developmental Pediatrician, Neurologist). When possible, diagnosis will be confirmed through the Children's Hospital of Philadelphia (CHOP) Electronic Health Record (EHR).
* Must identify an important person who is able to communicate by understanding and speaking full sentences in English
* Ability to communicate by understanding and using full sentences in English
* Informed Consent
* Be willing to have sessions audio- and video-recorded

Exclusion Criteria for Autistic Teens and Young Adults:

* Diagnosis of Intellectual Disability
* Participant is currently considered a suicide risk in the opinion of the Investigator or is currently demonstrating active suicidal or homicidal ideation or self-injurious behavior.
* Current, comorbid psychiatric disorder with sufficiently intense symptoms in the opinion of the Investigator that these symptoms may confound treatment.
* Changes to mental health treatment plan (ex. starting or ending therapy or psychotropic medications over the course of this intervention).
* Participation in a prior trial of our intrinsic motivation condition

Inclusion Criteria for Important Person:

* Age 18 years or older
* Must attend at least 15 minutes of each treatment session
* Ability to communicate by understanding and using full sentences in English
* Informed consent
* Be willing to have sessions audio- and video-recorded

Exclusion Criteria for Important Person:

- Is not willing to support the autistic teen/young adult with their daily living skill goal

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Motivation to Change | Up to 9 weeks.
  The primary outcome measure for this study is the individual's motivation to change and improve upon their daily living skill. Motivation will be measured through 4 separate questions that ask about one's desire, ability, need, and commitment to change. All 4 questions will use the same scale, which ranges from 1 - 10. A total score will be used as the measure. This total score will be calculated by adding the score from each individual question. A higher score indicates a greater level of motivation.

SECONDARY OUTCOMES:
Behavior Change Scale | Up to 9 weeks.
  The Behavior Change Scale is a one-question scale that was created by the study team. It asks how often the person completed their daily living skill goal over the past week with 4 response options: is not able to (0), never or almost never when needed (1), sometimes when needed (2), and always or almost always when needed (3). Each response option has a number associated with it and scores will be calculated based on that number. A higher score indicates a greater level of behavior change.
Empowerment Measure | Up to 9 weeks.
  This questionnaire measures a participant's level of empowerment by asking them to answer questions about different aspects of doing their daily living skill goal. For example, how much control they have over doing their goal, their opportunities for pursuing and taking the lead in doing their goal, and how capable they think they are. This questionnaire has 14 items and participants are asked to rate how much they agree or disagree on a 7-point scale. Higher scores indicate higher levels of empowerment.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin E Yerys, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- CHOP Center for Advanced Behavioral Healthcare, Philadelphia, Pennsylvania, United States